CLINICAL TRIAL: NCT01526577
Title: A Dose Blocked-randomized, Double-blind, Active and Placebo Controlled, Single and Multiple Dosing, Dose-escalation Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics and Food Effect
Brief Title: Study of LC23-1306 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LG-PYCL001; LC23-1306 (Other: LGLS)
Record Dates: First submitted 2012-01-20; First posted 2012-02-06 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2013-08

CONDITIONS: Acute Coronary Syndrome
Keywords: phase1; healthy subjects; antiplatelet agent
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Platelet Aggregation Inhibitors; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LC23-1306 (Experimental): experimental drug
  Interventions: Drug: LC23-1306
- placebo (Placebo Comparator): LC23-1306 placebo
  Interventions: Drug: placebo
- Ticagrelor (Active Comparator): active comparator
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: LC23-1306 — LC23-1306 10, 30, 100, 200, 400, 600 mg Placebo 10, 30, 100, 200, 400, 600 mg
  Other Names: antiplatelet agent
  Arms: LC23-1306
Drug: placebo — LC23-1306 placebo
  Arms: placebo
Drug: Ticagrelor — Ticagrelor 90mg
  Arms: Ticagrelor

SUMMARY:
This will be a dose block-randomized, double-blind, active and placebo controlled, single and multiple dosing, dose-escalation study to evaluate tolerability, safety and pharmacokinetic/pharmacodynamic characteristics. Adverse events, physical examinations, vital signs, ECG and laboratory tests will be conducted for safety/tolerability evaluation and serial blood samples and urine collections for pharmacokinetic and pharmacodynamic evaluations will be conducted at specified time points.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 50 years at screening
2. Subjects with Body Mass Index (BMI) between 18.0 (inclusive) and 27.0 kg/m2 (exclusive); and a total body weight between 55 kg (inclusive) and 90 kg (exclusive). BMI (kg/m2) = body weight (kg)/ {height (m)}2.
3. Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures.
4. Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Recruitment location: Seoul University Hospital
  * Recruitment period:
    * Single dose study recruitment period: 12Mar2012 ~ 18Sep2012
    * Muti-dose study recruitment period: 02Dec2012 ~ 05Aug2013
Pre-assignment Details: The subjects were enrolled in single dose study and multiple study separately. The subject enrolled in single dose study was not allowed to be enrolled in multiple dose study.
Groups:
- Single Dosing LC23-1306: experimental drug LC23-1306 10, 30, 100, 200, 400, 600 mg
- Multiple Dosing LC23-1306: LC23-1306 100, 200, 400, 600mg
- Multiple Dosing Ticagrelor 90mg: Active comparator
Period: Overall Study
Arm/Group | Single Dosing LC23-1306 | Single Dosing Placebo | Multiple Dosing LC23-1306 | Multiple Dosing Placebo | Multiple Dosing Ticagrelor 90mg
Started | 49 (1 more subject enrolled as a substitute for 1 withdrawn subject before the administration.) | 12 | 33 (1 more subject enrolled as a substitute for 1 withdrawn subject before the administration.) | 9 (1 more subject enrolled as a substitute for 1 withdrawn subject before the administration.) | 10 (2 more subjects were enrolled as the substitutes for 2 withdrawn subjects before the administration.)
Completed | 48 | 12 | 32 | 8 | 8
Not Completed | 1 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Multiple Dosing LC23-1306: Experimental drug LC23-1306 100, 200, 400, 600mg
- Total: Total of all reporting groups
Arm/Group | Single Dosing LC23-1306 | Single Dosing Placebo | Multiple Dosing LC23-1306 | Multiple Dosing Placebo | Multiple Dosing Ticagrelor 90mg | Total
Number analyzed (Participants) | 49 | 12 | 33 | 9 | 10 | 113
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 27 (4) | 27 (3) | 28 (4) | 26 (4) | 31 (6) | 27 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 49 | 12 | 33 | 9 | 10 | 113

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events of LC23-1306
Time Frame: 7 days (plus or minus 1 day)
Reporting Status: Not Posted

2. Primary Outcome: Pharmacodynamic Measurement
Description: Inhibition of platelet aggregation (IPA) was analized by the platelet aggregation test.
  * Among the time points that platelet aggregation rate was meausred, the result only at 8h post dosing was provided in result section.
Time Frame: 1D 0, 2, 8, 24h for single dose study / 1D and 7D 0, 2, 8, 12, 24h for multiple dose study
Measure: Number; unit: percentage of platelet inhibition
Arm/Group | LC23-1306 | Placebo | Ticagrelor
Number analyzed (Participants) | 80 | 20 | 8
percentage of platelet inhibition | 70 | 30 | 91.9

3. Secondary Outcome: AUC
Time Frame: pre-dose, up to 3 days post-dose
Reporting Status: Not Posted

4. Primary Outcome: Platelet Aggregation Test, Bleeding Test
Time Frame: pre-dose, up to 1 day post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- LC23-1306: Test drug.
- Ticagrelar: Active comparator
Arm/Group | LC23-1306 | Ticagrelar | Placebo
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/10 | 0/21
Other Adverse Events (participants affected / at risk) | 43/82 | 10/10 | 8/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LC23-1306 (N=82) | Ticagrelar (N=10) | Placebo (N=21)
Nausea and so on. (Gastrointestinal disorders) | 43 (50) | 10 (13) | 8 (8) — One of the related AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No